CLINICAL TRIAL: NCT00787618
Title: A Single-Dose, Open-Label, Parallel Group Study To Evaluate The Pharmacokinetics And Safety Profile Of PROELLEX® (CDB-4124) In Female Subjects With Various Stages Of Impaired Renal Function And In Healthy Female Volunteers
Brief Title: Evaluate PK and Safety of Proellex® in Females With Various Stages of Impaired Renal Function and Healthy Females
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Increased LFTs
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: ZP-006
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Results first posted 2014-08-25 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Renal Impairment
Keywords: Renal impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — telapristone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 50 mg Proellex Mild impairment (Active Comparator): 50 mg Proellex single dose Female subjects with mild renal impairment function.
  Interventions: Drug: 50 mg Proellex
- 50 mg Proellex Moderate (Active Comparator): 50 mg Proellex, Female subjects with moderate renal impairment function.
  Interventions: Drug: 50 mg Proellex
- 50 mg Proellex, Normal (Active Comparator): 50 mg Proellex, Female subjects with normal renal function.
  Interventions: Drug: 50 mg Proellex

INTERVENTIONS:
Drug: 50 mg Proellex — Single dose
  Other Names: Telapristone acetate; Proellex

SUMMARY:
PK and safety profile of Proellex® in females with various stages of impaired renal function

DETAILED DESCRIPTION:
The study will evaluate the pharmacokinetics and safety profile of Proellex® in females with various stages of impaired renal function and in volunteers with normal renal function

ELIGIBILITY:
Inclusion Criteria:

* Speak, read, and understand English or Spanish and is willing and able to provide written informed consent on an IRB-approved form prior to the initiation of any study procedures;
* Female, between the ages of 18 and 48 years with Body Mass Index (BMI) between 18 and 39, inclusive, is preferred
* Subject must meet the criteria of mildly or moderately impaired renal function or have normal renal function
* Subject with renal impairment must have evidence of stable disease
* If on medications for treatment of the complications of renal disease, and other concommitant chronic illnesses, subject must have been taking the medications at a stable dose for at least 10 days prior to the first Proellex® dosing date and are then to be continued at the same dose for the duration of the study.
* Negative urine pregnancy test at screening visit
* Subject must agree to use a medically acceptable and effective non-hormonal double barrier method of birth control
* Healthy subject must have no significant abnormal findings at the screening physical examination
* Subject is willing to remain in the clinic for the screening visit (approximately 1 day for the first screening visit) and for the treatment visit (approximately 3 days)
* Additional inclusion criteria may apply

Exclusion Criteria:

* Abnormal screening visit vital signs or clinical laboratory evaluation considered clinically significant
* Subject with clinically significant abnormal liver function
* Pregnant or lactating females, or women who are attempting or expecting to become pregnant at any time during the study or one month after the study
* An acute illness within five (5) days of study medication administration
* Subject with diagnosed or suspected carcinoma of the breast, reproductive organs or any other organ system
* Additional exclusion criteria may apply

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre van As, MD, PhD, Study Director — Repros Therapeutics Inc.
Locations (4):
- United States (4):
  - Clinical Pharmacology of Miami, Inc, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota
  - New Orleans Center for Clinical Research - Knoxville, Knoxville, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 50 mg Proellex Mild Impairment | 50 mg Proellex Moderate | 50 mg Proellex, Normal
Started | 3 | 0 | 3
Completed | 3 | 0 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study prematurely terminated, no data available
Groups:
- Total: Total of all reporting groups
Arm/Group | 50 mg Proellex Mild Impairment | 50 mg Proellex Moderate | 50 mg Proellex, Normal | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants]
Sex: Female, Male [Count of Participants; unit: Participants]
Region of Enrollment [Number; unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Proellex
Time Frame: 48 hours
Population: Study prematurely terminated
Arm/Group | 50 mg Proellex Mild Impairment | 50 mg Proellex Moderate | 50 mg Proellex, Normal
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: No adverse event data is available
Arm/Group | 50 mg Proellex Mild Impairment | 50 mg Proellex Moderate | 50 mg Proellex, Normal
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was prematurely terminated for safety reasons (Proellex studies were put on clinical hold due to liver toxicity). Sponsor was unable to pay vendor, and was therefore not provided with any study data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights